

## Phase 1, Online Only: Informed Consent for Surveys 09/20/2020

Jon M. Houck, Ph.D., and his associates from the Mind Research Network, is conducting a research project. The purpose of the research is to find out about how COVID-19 is affecting people and their use of alcohol. You are being asked to participate because you are an adult who drinks alcohol above the low-risk level.

Your participation will involve completing an online survey and a computer game where you inflate a balloon on your screen. The survey and game should take about 30 minutes to complete. The survey includes questions such as "How worried have you been about coronavirus", "Over the last 2 weeks, how often have you been bothered by feeling nervous, anxious, or on edge?" and "How much and for how long did you typically drink in a week during the past 30 days?". We will also ask whether and when you would be interested in participating in Phase 2, the in-person portion of this study.

Your involvement in the research is voluntary, and you may choose not to participate. You can refuse to answer any of the questions at any time. There are no known risks in this research, but some individuals may experience discomfort or loss of privacy when answering questions. All of the information we collect about you will be coded with a special study code number and will be kept on password protected computers, and stored securely in restricted and protected databases. All identifiable information (e.g., your name, date of birth) will be removed from the information collected in this project. After we remove all identifiers, the information may be used for future research or shared with other researchers without your additional informed consent.

You will be compensated \$20 for the time and inconvenience of participating in this study. If you provided inaccurate screening information, we will not be able to compensate you. If you think you may have provided inaccurate screening information, please contact us so that we can update your screening information. Please be sure to provide your current contact information when you take the survey. If we are not able to reach you, we will not be able to send your compensation. If we have questions about any of your answers to the survey, we may contact you to verify your answers before we send your compensation. If we are not able to reach you with these questions, we will not be able to send your compensation.

The findings from this phase of the project will provide information on how the coronavirus may affect people's drinking patterns and their well-being. If published, results will be presented in summary form only.

If you have any questions, concerns, or complaints about the research, please feel free to call the Principal Investigator, Jon M. Houck, at (505) 272-2869. If you have questions regarding your rights as a research participant, or about what you should do in case of any harm to you, or if you want to obtain information or offer input, please contact the UNM Office of the IRB (OIRB) at (505) 277-2644 or irb.unm.edu.

By clicking "I Agree" you will be agreeing to participate in the above described research.

| <ul><li>1. O I agree and consent (please complete and sign</li><li>O I do not agree or consent</li></ul> | n below) |
|---|---|
| 2. What is your first name? | |
| 3. What is your last name? | |
| 4. Please click the Add Signature link to the right to sign the consent. When you have finished, please click the "Next page" button below to go to the next page and finalize your | |
| consent. | Add Signature |

On the next page you will be able to view your consent form. When you have finished, please click the checkbox to certify your response. After you click the box and click the "Submit" button, you will be able to download a copy of your signed consent form.

| I certify that all the information in the document above is correct. I understand that clicking 'Submit' will electronically sign the form and that signing this form electronically is the equivalent of signing a physical document. |
|---|